CLINICAL TRIAL: NCT06340035
Title: Ultrasound Guided Peripheral Nerve Stimulation of Gluteal Nerves to Enhance Strength and Power in Individuals With Chronic Knee Pain: A Randomized Controlled Pilot Study
Brief Title: Percutaneous Peripheral Nerve Stimulation of Gluteus Nerves to Improve Hip Strength and Power
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Xavier Picañol Parraga, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20230901
Record Dates: First submitted 2024-03-17; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Chronic Pain; Chronic Knee Pain
Keywords: Peripheral Nerve Stimulation; TENS; Strength; Pain; Knee Pain; Rehabilitation; Neuromodulation
MeSH Terms: conditions — Chronic Pain; Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: This pilot study utilizes a randomized parallel-group design, focusing on procedure feasibility for future clinical trials, in line with extended CONSORT guidelines for pilot studies. Participants, selected through a convenience sampling method due to their chronic knee pain, received pre- and post-treatment evaluations to assess the effect on gluteal muscle function. Post-informed consent, participants were allocated to either TENS or ultrasound-guided percutaneous nerve stimulation via a computer-generated randomization process executed with GraphPad Software (San Diego, CA, USA), ensuring a balanced 1:1 ratio.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: In the study, blinding will be implemented to minimize bias. The evaluating clinician will be blinded to participant group assignments, ensuring assessments are unbiased. Similarly, the data analyst will also be blinded, analyzing data without knowledge of group allocations to maintain impartiality. Data will be handled objectively, with statistical methods applied blindly to compare treatment groups. Despite challenges in completely blinding participants due to the distinct nature of interventions, every effort will be made to minimize potential bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous Peripheral Nerve Stimulation (Experimental): Nerves are localized at an ultrasound-guided level and with respect to the vascular-nervous package two acupuncture needles are inserted, one for each nerve. The stimulation is the same as the TENS group: 10 stimulations x 10 times x 10 seconds, evoking the maximum contraction without pain.
  Interventions: Other: Percutaneous Peripheral Nerve Stimulation
- Transcutaneous electrical nerve stimulation (Active Comparator): Two surface electrodes are inserted at the level of the superior gluteal and inferior gluteal nerve tract. A protocol of 10 stimulations x 10 seconds of stimulations x 10 times is performed with a 10 second rest between each repetition. A maximum contraction evoked without pain is sought.
  Interventions: Other: TENS

INTERVENTIONS:
Other: TENS — The TENS group is subjected to transcutaneous current. Two surface electrodes are inserted at the level of the superior gluteal and inferior gluteal nerve tract. A protocol of 10 stimulations x 10 seconds of stimulations x 10 times is performed with a 10 second rest between each repetition. A maximum contraction evoked without pain is sought.
  Arms: Transcutaneous electrical nerve stimulation
Other: Percutaneous Peripheral Nerve Stimulation — In the pPNS group, the superior gluteal nerve and inferior gluteal nerve are stimulated percutaneously. The nerves are localized at an ultrasound-guided level and with respect to the vascular-nervous package two acupuncture needles are inserted, one for each nerve. The stimulation is the same as the TENS group: 10 stimulations x 10 times x 10 seconds, evoking the maximum contraction without pain.
  Arms: Percutaneous Peripheral Nerve Stimulation

SUMMARY:
The goal of this pilot clinical trial is to evaluate whether the ultrasound-guided percutaneous peripheral nerve stimulation through a needle results in greater gains in strength and power compared to the administration of current through surface electrodes in patients undergoing strength and power assessments. The main questions it aims to answer are:

Does percutaneous stimulation of the superior and inferior gluteal nerves using ultrasound-guided needles enhance strength and power more effectively than transcutaneous stimulation through electrodes?

Is the effectiveness of current delivery significantly different between percutaneous and transcutaneous methods when assessed with a linear encoder in a standarized hip extension exercise?

Participants will:

Be randomized into two groups: one undergoing ultrasound-guided percutaneous stimulation of the gluteal nerves (experimental group) and the other undergoing transcutaneous stimulation through electrodes (control group).

The same stimulation protocol at 10 Hz frequency with the maximum muscle contraction evoked without pain will be performed in both groups. Then, the participants will undergo strength and power assessment before and after therapy administration using a linear encoder in a hip extension exercise.

Researchers will compare the experimental group to the control group to see if the method of current delivery (percutaneous vs. transcutaneous) has a significant impact on the gains in strength and power. This comparison is based on the hypothesis that percutaneous delivery of current, guided by ultrasound, is more effective than simply positioning a surface electrode for transcutaneous stimulation. The evaluation of strength and power will be performed through a linear encoder that measures peak strength and concentric power in each repetition, conducted by a blind operator unaware of the patients' group allocations.

DETAILED DESCRIPTION:
This study delves into the comparative efficacy of two modalities of nerve stimulation for enhancing muscular strength and power: the percutaneous application of electrical current via acupuncture needles versus traditional transcutaneous electrical nerve stimulation (TENS). The overarching objective is to discern whether percutaneous peripheral nerve stimulation (pPNS), guided by ultrasound, facilitates superior gains in muscle strength and power in the gluteal muscles compared to conventional TENS.

Participants, suffering from chronic knee pain, were systematically randomized into two cohorts: the experimental group underwent ultrasound-guided pPNS targeting the superior and inferior gluteal nerves, whereas the control group received TENS. The experimental setup was meticulously designed to ensure the sole variable of distinction between groups was the method of electrical stimulation applied. pPNS was delivered using a biphasic asymmetric electric current, set to a frequency of 10 Hz, a pulse width of 240 microseconds, and an intensity tailored to achieve maximal muscle contraction without inducing pain, based on a protocol of ten 10-second stimulations interspersed with 10-second rest periods. This regimen was predicated on prior findings demonstrating its efficacy in augmenting isometric strength following femoral nerve stimulation. The control group was subjected to a parallel protocol, differing only in the application technique, wherein electrodes replaced needles, adhering to the same stimulation parameters.

The therapeutic efficacy of both interventions was assessed through a rigorous evaluation of strength and power before and after the administration of therapy. This assessment employed a linear encoder to measure peak strength and concentric power during the Hip Thrust exercise, a method chosen for its reliability in quantifying these parameters. The procedure entailed performing the exercise under three different loads (30%, 50%, and 70% of the participant's maximum capacity, 1RM), with the evaluation aimed at capturing the concentric peak power in each repetition until a noticeable decline in performance was observed.

The hypothesis posits that pPNS, by virtue of its targeted and invasive nature, will yield greater improvements in muscle strength and power than TENS, attributed to its more direct stimulation of the nerve fibers and the encompassing muscle groups. The underpinning rationale is that pPNS's ultrasound-guided approach allows for a more precise delivery of electrical current to the nerves, potentially overcoming limitations associated with the superficial and diffuse application of TENS.

For the analysis of the collected data, an initial evaluation of distribution characteristics will be performed utilizing visual tools such as Q-Q plots and density plots, complemented by statistical measures of kurtosis and skewness to understand the data's underlying structure. The Shapiro-Wilk test will be applied to assess the normality of residuals, ensuring the validity of subsequent statistical tests. Descriptive statistics, including the mean, median, mode, and standard deviation of the collected quantitative measures, will be thoroughly examined to summarize the data effectively. Additionally, the homogeneity of these variables across the dataset will be scrutinized.

Regarding inferential statistics, an exploratory approach will be adopted to estimate confidence intervals and discern trends in the data, particularly focusing on pre- and post-treatment differences both within individual subjects and between the groups. Due to the anticipation of non-normal data distribution and the structure of the study design (pretest-posttest control group), non-parametric statistical tests will be employed for the analysis. Specifically, the Mann-Whitney U test will facilitate between-group comparisons, while the Wilcoxon test will be used for related measurements to detect changes within groups over time.

Data analysis and visualization efforts will be supported by SPSS 23.0 software (SPSS Inc., IBM Chicago, IL, USA) and/or GraphPad Software (San Diego, CA, USA). For the interpretation of results, a 95% confidence interval and an alpha level of 0.05 will be established as thresholds for statistical significance. The creation of figures and graphical representations of the findings will be executed using Adobe Illustrator (San José, CA, USA), ensuring that the visual presentation of data is both clear and informative. This comprehensive approach to data analysis and visualization aims to elucidate the potential differences in efficacy between percutaneous peripheral nerve stimulation and transcutaneous electrical nerve stimulation in enhancing muscle strength and power, guiding future research and clinical applications in the field.

ELIGIBILITY:
Inclusion criteria:

* Adult athletes above the legal age threshold
* Amateur athletes
* Experiencing chronic knee pain
* Possessing a prior diagnosis related to their knee condition
* Competent in the execution of the hip thrust exercise

Exclusion criteria:

* Underage or elderly
* Significant co-existing medical conditions and/or comorbidities
* Professional athletes
* Sedentary lifestyle
* Lack of familiarity with the hip thrust exercise
* Needle phobia or rejection to peripheral stimulation techniques
* Considerable contraindications such as a history of knee surgery, current pregnancy, or issues related to blood clotting.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Hip Extension Concentric Peak Power (Watts) | Through study completion, 1 day
  This parameter quantifies the maximum power output a participant can generate during the concentric phase of a barbell hip thrust, performed at maximal velocity. The measurement is facilitated by a validated linear encoder system, ChronoJump, which captures motion data at a high sampling rate of 1000 Hz. This system translates the vertical displacement of the barbell and the execution time of the concentric phase into real-time power output. By integrating the bar's velocity with the mass being lifted.
Hip Extension Concentric Peak Strength (Newtons) | Through study completion, 1 day
  Real-time generated force, measured in newtons (N), is a pivotal outcome for assessing the impact of the interventions on the muscular strength during a hip extension exercise, specifically the barbell hip thrust performed at maximal velocity. This metric is derived using the ChronoJump linear encoder system, which accurately captures the motion and force exerted by the participant in real-time.

SECONDARY OUTCOMES:
Concentric Phase Velocity (m/s) | Through study completion, 1 day
  The velocity of movement execution, quantified in meters per second (m/s), is a parameter for evaluating athletic performance during strength exercises. It measures the speed at which an individual can complete the concentric phase of a lift, such as a barbell hip thrust. This velocity is indicative of the athlete's power and explosiveness.
Maximum Strength (1RM in kgs) | Through study completion, 1 day
  The one-repetition maximum (1RM) indirectly measured through the load-velocity profile incorporates three distinct points along the curve to estimate the maximum weight a participant can lift for a single repetition with maximal effort. This methodological approach leverages the relationship between the velocity of a lift and the load being moved, underpinning the premise that the speed at which a participant can perform an exercise decreases as the weight increases. By recording the velocity of the barbell at three different loads during the concentric phase of an exercise, such as the barbell hip thrust, and plotting these velocities against the respective weights, a linear or curvilinear relationship is established. This relationship is then extrapolated to determine the load corresponding to the theoretical velocity at which 1RM would occur.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Picañol Párraga, PhD(c), Principal Investigator — Hospital Clinic
Locations (1):
- University of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
In line with the commitment to share Individual Participant Data (IPD), the plan encompasses disseminating all collected IPD that underlie the results reported in a forthcoming scientific publication. This effort is designed to promote transparency and facilitate further research by providing comprehensive access to detailed datasets. To ensure adherence to ethical standards and protect participant privacy, all shared data will undergo an anonymization process.
Time Frame: Data will be available after the publication of the main results, allowing sufficient time for the primary research team to complete additional analyses.
Access Criteria: Access to the anonymized datasets will be granted upon request to researchers who provide a methodologically proposal.

REFERENCES:
- [Background] Gallego-Sendarrubias GM, Arias-Buria JL, Ubeda-D'Ocasar E, Hervas-Perez JP, Rubio-Palomino MA, Fernandez-de-Las-Penas C, Valera-Calero JA. Effects of Percutaneous Electrical Nerve Stimulation on Countermovement Jump and Squat Performance Speed in Male Soccer Players: A Pilot Randomized Clinical Trial. J Clin Med. 2021 Feb 10;10(4):690. doi: 10.3390/jcm10040690. PMID 33578911
- [Background] Beltra P, Ruiz-Del-Portal I, Ortega FJ, Valdesuso R, Delicado-Miralles M, Velasco E. Sensorimotor effects of plasticity-inducing percutaneous peripheral nerve stimulation protocols: a blinded, randomized clinical trial. Eur J Pain. 2022 May;26(5):1039-1055. doi: 10.1002/ejp.1928. Epub 2022 Mar 3. PMID 35191131
- [Background] de-la-Cruz-Torres B, Barrera-Garcia-Martin I, Romero-Morales C. Comparative Effects of One-Shot Electrical Stimulation on Performance of the Flexor Hallucis Longus Muscle in Professional Dancers: Percutaneous Versus Transcutaneous? Neuromodulation. 2020 Aug;23(6):865-870. doi: 10.1111/ner.13040. Epub 2019 Aug 25. PMID 31448488
- [Background] Requena Sanchez B, Padial Puche P, Gonzalez-Badillo JJ. Percutaneous electrical stimulation in strength training: an update. J Strength Cond Res. 2005 May;19(2):438-48. doi: 10.1519/13173.1. PMID 15903388
- [Background] Zhou S, Huang LP, Liu J, Yu JH, Tian Q, Cao LJ. Bilateral effects of 6 weeks' unilateral acupuncture and electroacupuncture on ankle dorsiflexors muscle strength: a pilot study. Arch Phys Med Rehabil. 2012 Jan;93(1):50-5. doi: 10.1016/j.apmr.2011.08.010. Epub 2011 Nov 8. PMID 22075372